CLINICAL TRIAL: NCT03870113
Title: Clinical Study on the Regress of Cervical Intraepithelial Neoplastic(CIN) 1/CIN2 by Highly Effective DC Vaccines Targeting HPV E6/ E7 Protein
Brief Title: DC Vaccines Targeting HPV16/18 E6/E7 Protein to Regress CINI/CIN2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShenzhenPH BTR-002
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical Intraepithelial Neoplasia; Human Papillomavirus; Dentritic Vaccine; E6/E7 protein
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccinated group (Experimental): Patients will be vaccinated with autologous mature dendritic cells-loaded with HPV 16/18 E6/E7, DC vaccine will be injected into the adjacent lymph-node 6 times, once a week.
  Interventions: Biological: Vaccinated group

INTERVENTIONS:
Biological: Vaccinated group — Develop highly reactive DC vaccines targeting HPV 16/18 E6/ E7 protein and DC vaccine would be injected to patients once a week, six doses in total.

SUMMARY:
To establish therapeutic dendritic cell (DC) vaccines targeting HPV 16/18 E6/E7 protein to block the progression of CIN1/CIN2 to cervical cancer and evaluate the safety and efficacy of the vaccines.

DETAILED DESCRIPTION:
Cervical cancer is the second most common cause of cancer-related deaths among women worldwide with 10000 new cases each year in China. The high-risk human papillomavirus (HPV) was the major cause of cervical cancer. The oncoproteins E6 and E7 encoded by HPV16 and 18, are consistently expressed in HPV-associated Cervical cancer and are responsible for the cervical cancer malignant progression. Targeting the E6/E7 proteins could be very helpful to regress the CIN 1/2 and block the tumorigenesis.

By this research, we aim to establish the HPV16/18 E6/E7 peptide library which could induce the strong anti-virus immune response and to vaccinate the CIN 1/2 patients with dendritic cell vaccines loaded HPV 16/18 E6/E7 epitopes.

Including:

1. To create an effective HPV 16/18 E6/E7 antigen peptide library using NetMHCspan software based on the MHC-I subtype of the Chinese population and screen E6/E7protein peptides with high binding affinity to MHC molecules;
2. To develop HPV 16/18 E6/E7- pulsed DC vaccines and evaluate the safety and efficacy of DC vaccines;
3. The patients are vaccinated with the HPV16/18 E6/E7- pulsed DC vaccines
4. To evaluate the safety and efficacy of DC vaccines loaded with HPV 16/18 E6/E7.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years ≤ 70 years at the time of informed consent
2. HPV type 16/18 positive
3. Pathologically confirmed CIN1/2 and no other cervical disease
4. adequate organ functions.

Exclusion Criteria:

1. Severe allergy to drugs
2. Women of child-bearing potential who are pregnant or breast-feeding
3. Any form of primary immunodeficiency
4. With serious cardiac, cerebrovascular and primary diseases
5. With a history of severe mental illness

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 3 months after the last vaccination injection
  Safety of personalized neoantigen vaccine will be measured by the number of subjects experiencing each type of adverse event. Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.
Immunogenicity of neoantigen-primed DC Vaccines | once per three month
  Immunogenicity of the DC vaccine will be measured to detect changes of neoantigen-specific T cells by flow cytometry.

SECONDARY OUTCOMES:
Objective Response Rate | once per three month
  Objective Response Rate will be measured by detection of protein expression of HPV E6 / E7and evaluation of CIN phase

CONTACTS AND LOCATIONS:
Overall Officials: Hui Qi, M.D., Study Director — Shen Zhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No